CLINICAL TRIAL: NCT01313416
Title: A Pilot Study to Test the Feasibility of the Combination of Gemcitabine and Anti-PD1 Monoclonal Antibody (CT-011) in the Treatment of Resected Pancreatic Cancer
Brief Title: Gemcitabine and CT-011 for Resected Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug supply issues
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Samir N. Khleif, Cancer Center Director, Augusta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-C-0100
Record Dates: First submitted 2011-03-10; First posted 2011-03-11 (Estimated); Results first posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-06

CONDITIONS: Pancreatic Neoplasms; Cancer of the Pancreas; Neoplasms Pancreatic; Pancreatic Cancer; Pancreas Cancer
Keywords: Adjuvant Therapy; Recombinant Monoclonal Antibody; Adenocarcinoma of the Pancreas; Vaccination; PD-1 Receptor; Pancreas Cancer; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — pidilizumab; spartalizumab; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Experimental): Combination CT-011 and Gemcitabine
  Interventions: Biological: CT-011; Drug: Gemcitabine

INTERVENTIONS:
Biological: CT-011 — 3mg/kg, intravenous (IV) day 1 of each cycle over 2 hours.
  Other Names: Anti-PD1 Antibody
Drug: Gemcitabine — 1000mg/m^2 intravenous (IV) over 30 minutes on days 8, 15, and 22 of each cycle.
  Other Names: Gemzar

SUMMARY:
Background:

* In 2009, 49,096 patients were diagnosed with pancreatic cancer. Pancreatic cancer carries a poor prognosis with an overall 5-year relative survival rate of 5.6%.
* Many doctors believe that individuals who have had surgery to remove pancreatic cancer should receive additional treatment, known as adjuvant therapy or adjuvant treatment, to prevent the cancer from returning. One chemotherapy drug that has been found to be effective in some patients with pancreatic cancer is called gemcitabine; it has been shown to improve patient survival by 6 months. Researchers are searching for new drugs or drug combinations to improve on these results.
* One of the leading causes for immune suppression in cancer patients was suggested to be associated with the elevated expression of programmed cell death ligand 1 (PD-L1) human B7 homolog 1 (B7-H1) at tumor-involved sites, either by the tumor itself or by surrounding cells like regulatory immune cells, resulting in the local suppression and apoptosis of tumor infiltrating effector lymphocytes.
* Some chemotherapy drugs kill cancer cells directly, but appear to prevent the immune system from helping in that fight. The experimental drug CT-011 is designed to help the immune system remain active to fight cancer cells. CT-011 has been tested in laboratories and studied for use with a number of other cancers, but it has not been given in combination with gemcitabine as a treatment for pancreatic cancer.

Objective:

- To test the safety and effectiveness of chemotherapy drugs gemcitabine and CT-011 as a follow-up treatment for pancreatic cancer that has been surgically removed.

Eligibility:

- Individuals at least 18 years of age who have had surgery to remove pancreatic cancer and have not had other types of follow-up treatments.

Design:

* Participants will receive gemcitabine and CT-011 in 28-day cycles of treatment, and will be monitored throughout their treatment.
* Participants who do not have serious side effects and remain cancer-free may receive this drug combination every 28 days for a total of 6 cycles.
* Participants will have follow-up visits with additional blood tests every 2 months after stopping treatment for up to 2 years.

DETAILED DESCRIPTION:
RATIONALE:

* CT-011 is a humanized immunoglobulin G 1 (IgG1) kappa recombinant monoclonal antibody against PD-1 receptor that blocks the interaction of PD-L1 with PD-1. CT-011 specifically binds to an epitope that is shared between the murine and the human PD-1 receptors on activated T cells, B cells, natural killer (NK) cells, and myeloid cells (CD14+ cells) and primarily functions in effector/memory T lymphocytes and in NK cells. In a functional bioassay, CT-011 was demonstrated to block the activity of PD-1 and to operate on CD4+CD45RO+ effector/memory T lymphocytes leading to attenuation of apoptotic processes.
* CT-011 was studied in experimental murine tumor models of melanoma, lung cancer, fibrosarcoma, leukemia/lymphoma and colorectal carcinoma and was shown to inhibit tumor growth and extend the survival of tumor-bearing nude mice, and to generate tumor-specific protection against tumor re-challenge.
* Recent findings have demonstrated that chemotherapies like paclitaxel, etoposide or fluorouracil (5-FU) induce the expression of the PD-L1 on tumor cell lines leading to an immune-suppressive environment and promoting PD-L1-mediated T cell apoptosis

The study will be conducted as an optimal two-stage phase II trial, in order to rule out an unacceptably low 50% of patients who do not receive the full dose of CT-011 (p0=0.50) in favor of a modestly high 80% fraction who receive the full dose of CT-011 (p1=0.80). It is anticipated that up to 32 patients may be enrolled onto this trial.

OBJECTIVES:

* Primary endpoint: To determine the feasibility and safety of the combination of CT-011 and Gemcitabine in patients after primary macroscopic resection of pancreatic carcinoma.
* Secondary endpoint: To determine if the addition of CT-011 to Gemcitabine can improve the median disease-free survival in resected pancreatic cancer.

DESIGN:

* Eligible subjects will be screened with a full medical history and physical examination, blood and urine tests, and imaging studies.
* Participants will receive adjuvant combination CT-011 and Gemcitabine in 28-day cycles.
* CT-011 will be given at a dose of 3mg/kg by intravenous infusion over 2 hours on day 1, one week prior to the first Gemcitabine infusion of each cycle.
* Gemcitabine will be given at a dose of 1000mg/m^2 by intravenous infusion over 30 minutes on Days 8, 15 and 22 of each cycle.
* Treatment will be continued for a total of 6 cycles or until disease recurrence or grade IV non-hematological toxicity if occurred before the completion of 6 cycles.
* Participants will be monitored with frequent blood and urine tests throughout their treatment visits. Every other cycle (about every 2 months), participants will also have imaging studies to evaluate the experimental treatment.
* Participants will have follow-up visits with additional blood tests every 2 months after stopping treatment for up to 2 years.

ELIGIBILITY:
* Adult patients with histologic verification of carcinoma of the pancreas (T1-3, N0-1) who have undergone surgical resection within the past 4 - 12 weeks. Patients with R1 resections are excluded.
* Must meet all laboratory safety criteria and not have active or history of autoimmune disease or conditions, be treated with immunosuppressive drugs, or require the use of systemic steroids. Primary intraoperative chemotherapy will be allowed.
* Pregnant or nursing women will be excluded. Subjects with active infection, HIV, Hepatitis B or C will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir N. Khleif, MD, Principal Investigator — Augusta University
Locations (1):
- Georgia Regents University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
Comprehensive data will be reported, not individual participant data.

REFERENCES:
- [Background] Geer RJ, Brennan MF. Prognostic indicators for survival after resection of pancreatic adenocarcinoma. Am J Surg. 1993 Jan;165(1):68-72; discussion 72-3. doi: 10.1016/s0002-9610(05)80406-4. PMID 8380315
- [Background] Sener SF, Fremgen A, Menck HR, Winchester DP. Pancreatic cancer: a report of treatment and survival trends for 100,313 patients diagnosed from 1985-1995, using the National Cancer Database. J Am Coll Surg. 1999 Jul;189(1):1-7. doi: 10.1016/s1072-7515(99)00075-7. PMID 10401733
- [Background] Saif MW. Adjuvant treatment of pancreatic cancer in 2009: where are we? Highlights from the 45th ASCO annual meeting. Orlando, FL, USA. May 29-June 2, 2009. JOP. 2009 Jul 6;10(4):373-7. PMID 19581737
- [Background] Miller RC, Iott MJ, Corsini MM. Review of adjuvant radiochemotherapy for resected pancreatic cancer and results from Mayo Clinic for the 5th JUCTS symposium. Int J Radiat Oncol Biol Phys. 2009 Oct 1;75(2):364-8. doi: 10.1016/j.ijrobp.2008.11.069. PMID 19735864

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Toxicity Evaluation: From Time of First Treatment With CT-011 (Pidilizumab, MDV9300)
Description: Patients presenting with symptoms possibly related to autoimmune reaction will be evaluated for organ specific autoimmune involvement, i.e:
  * Acute abdominal symptoms should be evaluated for pancreatitis, including lipase and amylase levels;
  * Persistent diarrhea should be evaluated for infection (c. diff). Any suspicion of colitis should be evaluated by a colonoscopy with biopsy.
  * Visual symptoms should be immediately evaluated by an ophthalmologist.
  * Generalized rash should be biopsied prior to local skin care, antihistamines or corticosteroids.
  * Pulmonary symptoms will be evaluated immediately, including repeated PFTs (pulmonary function tests).
Time Frame: 2 years
Population: Study discontinued due to drug supply issues prior to analysis; no meaningful data derived.
Arm/Group | Single Arm
Number analyzed (Participants) | 0

2. Secondary Outcome: Disease Response: Evaluated Using the Revised Response Evaluation Criteria in Solid Tumors (RECIST) Guidelines (v1.1)
Description: Patients who have received at least one cycle of therapy will be evaluated for response every 8 weeks (every other cycle). Confirmatory scans will be obtained 4 weeks following initial documentation of objective or non-target disease response.
  Response will be evaluated on target and non-target lesions. The same method of assessment and same technique will be used to characterize each identified and reported lesion at baseline and during follow-up. Response will be reported as:
  * Complete Response (CR); Disappearance of all target lesions
  * Partial Response (PR); At least 30% decrease in the sum of the diameters of target lesions
  * Progressive Disease (PD): At least 20% increase in the sum of the diameters of target lesions. The sum must also demonstrate an absolute increase of at least 5 mm.
  * Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: 2 years
Population: Study discontinued due to drug supply issues prior to analysis; no meaningful data derived.
Arm/Group | Single Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Single Arm
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other